CLINICAL TRIAL: NCT06269289
Title: Effects of Web-Based Education on Patient Empowerment and Asthma Control in Asthma Patients
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Saglik Bilimleri Universitesi (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: SBU-KOMSERN-001
Record Dates: First submitted 2024-02-12; First posted 2024-02-21 (Actual); Last update posted 2024-02-21 (Actual); Status verified 2024-02

CONDITIONS: Asthma; Patient Empowerment
Keywords: asthma; web based intervention; education; nursing; patient empowerment
MeSH Terms: conditions — Asthma; Patient Participation

STUDY DESIGN:
Intervention Model Description: The research was designed as a randomized controlled experimental study with a pretest-posttest design.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- intervention group (Experimental): It will be determined using a table of random numbers. The group has been diagnosed for at least 1 year, It will consist of people (25) between the ages of 18-65, who can read and write in Turkish, who volunteer to participate in the study and who have not received any training before. After meeting the individuals and obtaining their verbal and written consent, they will be asked to fill out the Patient Information Form, Patient Empowerment Scale and Asthma Control Test obtained through Google Forms. Post-tests will be applied to individuals who complete all 5 modules of training.
  Interventions: Other: web based education
- Control group (Active Comparator): The participants will be individuals who apply to the Allergy and Immunology Clinic of Istanbul Sureyyapasa Chest Diseases and Surgery Training and Research Hospital, have been diagnosed with asthma for at least one year and agree to participate in the study. It will consist of people who are between the ages of 18-65, understand Turkish, know how to read and write. Twenty five people selected by the randomization table method will be in the control group. They will be given the Ministry of Health's asthma education brochure. As in the intervention group, pre-test and post-test will be conducted.
  Interventions: Other: Standard education brochure

INTERVENTIONS:
Other: web based education — Training presentations will be prepared in 5 modules by taking expert opinions in line with the literature. Training will be aimed at empowering patients to control asthma. It will include topics such as medication use, device use, exercise and disease management. Each week, an intervention group will be invited online to a module and the training will be given by the researcher.
  Arms: intervention group
Other: Standard education brochure — The control group will not be given web-based training, but will be given the standard asthma education brochure of the Ministry of Health.
  Arms: Control group

SUMMARY:
Asthma is defined as a chronic inflammatory disorder of the airways associated with an extreme increase in airway hyperresponsiveness leading to recurrent wheezing, shortness of breath, chest tightness, and coughing attacks. The World Health Organization states that approximately 339 million individuals worldwide have asthma and more than 400 thousand deaths occur due to asthma every year.

With effective and sustainable asthma management, it is possible to reduce disease-related complaints, admissions to emergency units and hospitalizations, limit the physiological and psychological effects of the disease, prevent dependence on healthcare professionals and caregivers, increase the quality of life and reduce the mortality of the disease. Patient education, which is within the educational role of professional nurses, is very important in asthma management. The research was planned in a single-center, randomized control group pretest-posttest design. The sample will consist of individuals who applied to the Allergy and Immunology clinic of Sureyyapasa Chest Diseases and Surgery Training and Research Hospital between May 2024 and January 2024, who have been diagnosed with asthma for at least one year and who accept the study [25 intervention group - 25 control group]. Groups will be determined using the random numbers table from the simple random sampling method. A web-based asthma education module will be created in line with the literature, and participants in the intervention group will be given synchronous training in 5 modules. After meeting the individuals in the intervention and control groups and obtaining verbal and written consent, they will be asked to fill out the Patient Information Form, Patient Empowerment Scale and Asthma Control Test prepared via Google Forms. A 30-minute training session will be given to the intervention group every week and there will be short evaluations after each training. When the 5th Module is completed, the intervention group will be asked to fill out the Patient Empowerment Scale and Asthma Control Test Scale. No intervention will be applied to the control group. 5. At the end of the module, the Patient Empowerment Scale and Asthma Control Test will be completed by individuals in the control group. It is thought that web-based asthma education that individuals will receive will positively affect their empowerment levels and increase their disease control.

DETAILED DESCRIPTION:
The episodic nature of asthma symptoms and exacerbations makes effective self-management of the condition a necessity. Less than 40% of individuals with asthma monitor their symptoms regularly, and the proportion who initiate a prescribed course of action at the first sign of an exacerbation is even lower. Many patients have difficulty recognizing early signs of worsening and often fail to implement asthma action plans.

Many factors such as air pollution, genetic factors, cigarette smoke, allergens, respiratory infections and stress contribute to the development of asthma and triggering attacks. For this reason, a multifaceted approach is required in the treatment and control of asthma.

People with severe asthma may have debilitating symptoms that persist despite high-dose treatment. Clinical guidelines for severe asthma recommend concepts such as patient-centeredness, shared decision-making, and self-management, with autonomy at its core. To improve outcomes in individuals with mild or severe asthma, guidelines emphasize the importance of patient-centeredness, shared decision-making, and self-management. Central to these concepts is autonomy, a term widely used and valued in the healthcare literature for which there is no gold standard definition.

In parallel with the developments and changes in the field of information technology in recent years, the internet has replaced classical communication and teaching applications and has become used in many different areas such as keeping up with current information, social sharing, communicating professionally, shopping, banking transactions and education. Internet use has also become increasingly widespread in the field of health. Internet users can obtain ideas about their own health and the health of the individuals around them through the information they obtain from health websites.

Today, meeting the increasing demand for health services and supporting nursing care requires greater use of technology. Nurses who care for a healthy/sick individual and are closest to them should have all the information about the individuals' health as soon as possible in order to provide quality care, ensure their safety and interact quickly. Effectively used technology prevents waste of medical equipment, ensures proper use of resources, evidence-based practice, and improves standards and quality of care by providing clinical decision-making support. Nurses use technology as a tool of change by directing this process and policies in order to provide quality, qualified and low-cost care to individuals and society.

Web-based education (WTE), which is a distance education method, is defined as an education program created by taking advantage of the features of the internet and computer technologies.

Web-based training is classified as synchronous or asynchronous according to the communication method. Synchronous education is a method in which two-way communication is provided and mutual interaction occurs simultaneously, although the teacher and the student are physically in different environments.

WTE systems allow individuals to receive education independently of time, place and distance. WTE systems are widely used in the healthcare field, especially in the management of chronic diseases. This burden placed on the healthcare system by individuals with chronic diseases puts a strain on all countries of the world, including countries with strong social security systems; Many countries are turning to home care, which is a more economical system, instead of costly institutional care, the role of hospitals is limited to acute health care, and family members are expected to take a greater role in care.

Educational programs aimed at individuals, families and society aim to prevent diseases and improve health; There are many studies showing that it is effective in providing disease management for those who are sick. WTE programs are cost-effective because they can reach large audiences in a short time and save time.

Web-based self-care interventions have the potential to reduce health disparities by removing barriers to accessing health care. However, there is a lack of evidence on the effects of these interventions on chronic conditions.

The cornerstones of asthma treatment are guideline-based medication adherence and asthma education programs that aim to equip the individual for effective self-management of the disease.

ELIGIBILITY:
Inclusion Criteria:

* Receiving treatment with a diagnosis of asthma for at least 1 year
* Having severe asthma
* Not having had any previous training
* Being between the ages of 18-65,
* Knowing how to read, write,
* Volunteering to participate in research

Exclusion Criteria:

* Having received treatment for less than 1 year
* Being educated,
* Not being at the level of severe asthma,
* Not meeting the age criterion,
* Not having the ability to understand, read and write Turkish

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-05-30 (Estimated); Primary Completion 2024-06-30 (Estimated); Study Completion 2024-09-30 (Estimated)

PRIMARY OUTCOMES:
patient empowerment scale (PES) | five weeks
  The scale consists of 37 items and five factors. Scale rating: 5-point Likert (1 = strongly disagree - 5 = strongly agree) The score that can be obtained from the scale varies between 37 and 185. As the score from the scale increases towards 5, patient empowerment is considered high, and as it decreases towards 1, patient empowerment is considered low.

SECONDARY OUTCOMES:
Asthma Control Test (ACT) | five weeks
  A self-administered questionnaire containing five items assessing frequency of shortness of breath, general asthma symptoms, use of rescue medications, impact of asthma on daily functioning, and overall self-assessment of asthma control. Each item contains five response options with values ranging from 1 to 5. An ACT score of <20 indicates uncontrolled asthma.

CONTACTS AND LOCATIONS:
Overall Officials: Neslihan Komser, Principal Investigator — SUREYYAPASA CHEST DISEASES AND THORACIC SURGERY TRAINING AND RESEARCH HOSPITAL
Locations (1):
- Sureyyapasa Chest Diseases and Thoracic Surgery Training and Research Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No